CLINICAL TRIAL: NCT04092920
Title: Primary Implant Stability of Laser Surface Treated Versus Sand Blasted/Acid Etched Surface Treated Implants in Fresh Extraction Sockets: A Randomized Clinical Trial
Brief Title: Implant Stability of Laser vs SLA Surface Treated Implants Placed in Fresh Extraction Sockets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed mohamed mohamed abd el maksoud, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO 6-3-1
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Implant Site Reaction
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laser and SLA implants (Experimental): extraction of badly broken maxillary and mandibular teeth with immediate implant placement using laser surface treated and SLA surface treated dental implants
  Interventions: Device: laser and SLA

INTERVENTIONS:
Device: laser and SLA — ligible patients will be randomized to 2 groups control group will receive SLA surface treated implant to replace badly broken tooth immediately after extraction and a study group will receive laser surface treated implant to replace badly broken tooth immediately after extraction.
  atraumatic extraction will be performed and socket will be examined for presence of bone dehesince or fenestration if no, implant will be placed immediately and a implant primary stability will be measured using an ISQ unit and recorded as base Line reading .
  gingival former will be attached to the implant and removed at 2 ,4,8,12 week intervals to record ISQ readings.

SUMMARY:
Commercially available implant surfaces are moderately roughened surfaces and they are obtained by acid-etching following alumina or titanium oxide grit-blasting.

Although the micro-rough implants can be successful in compromised clinical scenarios, the bioinert nature of titanium surfaces cannot stimulate a more rapid bone regeneration and mechanical fixation of dental implants.

Laser surface treatment is used to produce an implant surface modification on the nano-scale with controlled and reproducible patterns in addition to exhibiting a sterilizing effect and achieving efficient oxidation .

DETAILED DESCRIPTION:
For dental implant to be successful, a direct contact between the bone tissue and the surface of the implant should be developed & this physiological phenomenon is known by the term of osseointegration.

Initially, it was supposed that to achieve osseointegration, implants had to be submerged under the mucosa & left without any loading for a period of 3-4 months in mandible and 6-8 months in maxilla.

Recently immediate implant placement at the time of extraction has become a viable treatment alternative, this approach provides the advantages of decreasing the patient's discomfort, the treatment's duration and costs.

Aiming to reduce healing process to limit such changes in the soft & hard tissues and reducing treatment time, several alterations in both surgical and restorative procedures has been introduced. From an implant design perspective, two approaches including the fields of biomaterials and/or biomechanics have been most utilized; implant body design which aim to increase the primary stability and surface modifications to allow faster osseointegration process.

Rough implant surface is modified by different techniques. Among these different techniques, interest in of using laser to achieve roughened surfaces.

Commercially available implant surfaces are moderately roughened surfaces and they are obtained by acid-etching following alumina or titanium oxide grit-blasting.

Although the micro-rough implants can be successful in compromised clinical scenarios, the bioinert nature of titanium surfaces cannot stimulate a more rapid bone regeneration and mechanical fixation of dental implants.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with badly broken teeth indicated for extraction. • Presence of adequate bone beyond the root apex to guarantee implant primary stability & implant placement within the alveoli confines.

Exclusion Criteria:

* • Presence of acute infections in the implant site.

  * Presence of fenestrations or dehiscence of the residual bony walls after extraction.
  * Heavy smokers more than 20 cigarettes per day.
  * Patients with systemic disease that may affect normal healing.
  * Psychiatric problems.
  * Disorders to implant are related to history of radiation therapy to the head and neck neoplasia.
  * Immunodeficiency pathology, bruxism, stress situation (socially or professionally), emotional instability, and unrealistic aesthetic demands.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
rate of change in implant stability at baseline,2,4,8,12 weeks | 3 months
  measuring implant stability with Resonance Frequency Analysis device using Implant stability quotient (ISQ) units that measure the stiffness and deflection of the implant-bone complex.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt